CLINICAL TRIAL: NCT00817128
Title: Pain Exposure Physical Therapy Or Conservative Therapy for Patients With Complex Regional Pain Syndrome Type I
Brief Title: Pain Exposure Physical Therapy (PEPT) Versus CBO in Patients With Complex Regional Pain Syndrome Type I (CRPS-1)
Acronym: PEPTOC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Jan Paul Frolke, MD PhD, Department of Surgery, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170991004; ZonMw 1709901004 (Other Grant/Funding Number: ZonMw 1709901004)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Complex Regional Pain Syndrome, Type I
Keywords: Complex Regional Pain Syndrome Type I; Sympathetic Reflex Dystrophy; Pain Exposure Physical Therapy; Pharmacological treatment; Functional recovery
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Complex Regional Pain Syndromes | interventions — 1,10-phenanthroline-platinum(II)-ethylenediamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PEPT after randomization
  Interventions: Procedure: PEPT
- 2 (Experimental): CBO after randomization
  Interventions: Procedure: CBO standard

INTERVENTIONS:
Procedure: PEPT — Pain Exposure Physical Therapy
  Arms: 1
Procedure: CBO standard — Standard therapy as defined in CBO guideline 2006
  Arms: 2

SUMMARY:
The current Dutch CBO guideline treatment of Complex Regional Pain Syndrome Type I (CRPS-1) is very disappointing with chronification, disability and subsequent high medical costs and personal suffering. A possible better treatment is intensive function-oriented physical therapy or Pain Exposure in Physical Therapy (PEPT). However, there are no adequate studies performed that demonstrate the efficacy of PEPT and therefore PEPT is lacking in the Dutch CBO CRPS-1 guidelines. Despite a lacking scientific argumentation, the PEPT approach or Macedonian therapy, is now being adopted on a large scale among physical therapists in The Netherlands. There are two level C retrospective cohort studies demonstrating a promising and clinical relevant beneficial effect on pain and function after PEPT. In response to the growing demand for scientific argumentation among doctors and physical therapists with respect to the efficacy of PEPT, we conducted a pilot study at the UMC St Radboud Nijmegen. The results of this pilot study were very promising and therefore, we decided to design a large RCT to investigate the treatment effects and costs in CRPS patients treated with PEPT compared to CRPS patients treated with usual therapy according to the Dutch CBO guidelines.

DETAILED DESCRIPTION:
Hypothesis:

PEPT is expected to be 30% more effective and around three-folds cheaper than usual therapy (CBO)

Objective:

The current Dutch CBO guideline treatment of Complex Regional Pain Syndrome Type I (CRPS-1) is very disappointing with chronification, disability and subsequent high medical costs and personal suffering. A possible better treatment is intensive function-oriented physical therapy or Pain Exposure in Physical Therapy (PEPT). However, there are no adequate studies performed that demonstrate the efficacy of PEPT and therefore PEPT is lacking in the Dutch CBO CRPS-1 guidelines. Despite a lacking scientific argumentation, the PEPT approach or Macedonian therapy, is now being adopted on a large scale among physical therapists in The Netherlands. There are two level C retrospective cohort studies demonstrating a promising and clinical relevant beneficial effect on pain and function after PEPT. In response to the growing demand for scientific argumentation among doctors and physical therapists with respect to the efficacy of PEPT, we conducted a pilot study at the UMC St Radboud Nijmegen. The results of this pilot study were very promising and therefore, we decided to design a large RCT to investigate the treatment effects and costs in CRPS patients treated with PEPT compared to CRPS patients treated with usual therapy according to the Dutch CBO guidelines.

Study design:

Prospective, single-blinded, randomized clinical trial. After base-line measurements (T0), measurements are performed at three (T1) and six months (T2) after inclusion. Follow-up is at nine months (T3).

Study population:

Patients with Complex Regional pain Syndrome (CRPS-1) of either upper or lower extremity according to Bruehl's/IASP criteria (see attachment) between 3 and 24 months after initial injury will be selected for the study. After information about standard and experimental treatments for CRPS and after informed consent, patients will enter the study and randomization for usual (CBO) or experimental (PEPT) treatment will be performed.

Intervention:

Treatment group: In the treatment group medication prescribed for CRPS is tapered to zero. No invasive treatments like sympathetic blocks, and/or operations will be performed. After information about the mechanism of action of PEPT in relation to CRPS, patients receive five sessions of PEPT including homework exercises. The basic of PEPT is a function-oriented exercise therapy. The PEPT physical therapist manipulates restricted joints and intensively trains functional skills irrespective of pain experience during or after the therapy. Patients are stimulated to use an active coping style to achieve a clear functional goal in 5 sessions.

Control group: Usual treatment of CRPS according to the Dutch CBO CRPS guideline 2006 including, analgesics (WHO pain ladder), neuropathic drugs, N-acetylcysteine, calcium channel blocker, ketanserin and DMSO (dimethylsulphoxide). On indication, percutaneous sympathetic blocks or spinal cord stimulation will be performed. In addition, patients receive physical therapy with exercises within pain limits (pain contingent), splints and if necessary, aids for ADL activities.

Outcome measures:

Primary outcome measure is the Impairment level SumScore (ISS), which consists of three measurement parameters (pain, active range of motion and temperature) and four measurement instruments (VAS, McGill Pain Questionnaire, goniometry of mobility of joints and skin thermometer). A cost-effectiveness analysis from a societal perspective comparing PEPT to usual care in patients with CRPS will be performed. This will be done along-side the clinical trial.

Sample size calculation/data analysis:

The sample size calculation is based on the following finding and expectation. The improvement in ISS (primary outcome) over one year for the standard physical therapy group was 50% [Oerlemans, APMR 2000], for the PEPT group it is estimated at minimal 70-80%. Given an alpha of 0,05 and a power of 80% for a one sided Chi-square test 31 patients are needed per group. The Student T- test is used to calculate differences between both groups in mean ISS.

ELIGIBILITY:
Inclusion Criteria:

Patients between 18 and 80 years of age with Complex Regional pain Syndrome (CRPS-1) of either upper or lower extremity according to Bruehl's/IASP criteria between 3 and 24 months after initial injury will be selected for the study.

Exclusion Criteria:

Patients who do not comply with the inclusion criteria especially those who have other causes that may explain a pain syndrome will be excluded (IASP criterium)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure is the Impairment level SumScore (ISS): pain, active range of motion and temperature, measured with VAS, McGill Pain Questionnaire, goniometry of mobility of joints and skin thermometer | t=0; t= 3 months; t= 6 months; t= 9 months

SECONDARY OUTCOMES:
DASH; FABQ; SF36; mycrofet dynamometer; RSQ; 10 meter walking test and the timed up-and-go-test; Adherence behavior; Seven Days PAR; IPAQ; PCS; PDI; PAM; Economic evaluation with diary; EuroQol 5D; adverse reactions SAE forms | t=0; t=3 months; t= 6 months; t= 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Frölke, MD; PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Background] Oerlemans HM, Oostendorp RA, de Boo T, van der Laan L, Severens JL, Goris JA. Adjuvant physical therapy versus occupational therapy in patients with reflex sympathetic dystrophy/complex regional pain syndrome type I. Arch Phys Med Rehabil. 2000 Jan;81(1):49-56. PMID 10638876
- [Background] Sherry DD, Wallace CA, Kelley C, Kidder M, Sapp L. Short- and long-term outcomes of children with complex regional pain syndrome type I treated with exercise therapy. Clin J Pain. 1999 Sep;15(3):218-23. doi: 10.1097/00002508-199909000-00009. PMID 10524475
- [Background] Perez RS, Oerlemans HM, Zuurmond WW, De Lange JJ. Impairment level SumScore for lower extremity Complex Regional Pain Syndrome type I. Disabil Rehabil. 2003 Sep 2;25(17):984-91. doi: 10.1080/0963828031000122302. PMID 12851087
- [Background] Vaneker M, Wilder-Smith OH, Schrombges P, Oerlemans HM. Impairments as measured by ISS do not greatly change between one and eight years after CRPS 1 diagnosis. Eur J Pain. 2006 Oct;10(7):639-44. doi: 10.1016/j.ejpain.2005.10.003. Epub 2005 Nov 21. PMID 16300975
- [Background] Frolke JP, Bruggeman AW, Klomp FP, Smeets JL. Brugada syndrome during physical therapy: a case report. Cases J. 2008 Aug 18;1(1):107. doi: 10.1186/1757-1626-1-107. PMID 18710557
- [Derived] Barnhoorn KJ, van de Meent H, van Dongen RT, Klomp FP, Groenewoud H, Samwel H, Nijhuis-van der Sanden MW, Frolke JP, Staal JB. Pain exposure physical therapy (PEPT) compared to conventional treatment in complex regional pain syndrome type 1: a randomised controlled trial. BMJ Open. 2015 Dec 1;5(12):e008283. doi: 10.1136/bmjopen-2015-008283. PMID 26628523
- [Derived] Barnhoorn KJ, Staal JB, van Dongen RT, Frolke JP, Klomp FP, van de Meent H, Samwel H, Nijhuis-van der Sanden MW. Are pain-related fears mediators for reducing disability and pain in patients with complex regional pain syndrome type 1? An explorative analysis on pain exposure physical therapy. PLoS One. 2015 Apr 28;10(4):e0123008. doi: 10.1371/journal.pone.0123008. eCollection 2014. PMID 25919011
- [Derived] Barnhoorn KJ, Oostendorp RA, van Dongen RT, Klomp FP, Samwel H, van der Wilt GJ, Adang E, Groenewoud H, van de Meent H, Frolke JP. The effectiveness and cost evaluation of pain exposure physical therapy and conventional therapy in patients with complex regional pain syndrome type 1. Rationale and design of a randomized controlled trial. BMC Musculoskelet Disord. 2012 Apr 19;13:58. doi: 10.1186/1471-2474-13-58. PMID 22515496